CLINICAL TRIAL: NCT07316062
Title: A Multi-centre Chart Review Study on the Treatment Patterns and Outcomes of Stage I-III Non-Small Cell Lung Cancer in China
Brief Title: A Multi-centre Chart Review Study of Stage I-III Non-Small Cell Lung Cancer in China
Acronym: MAP
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00236
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Non-Small-Cell Lung
Keywords: NSCLC, chart review
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This chart review study is proposed in China to understand the treatment patterns, biomarker testing, and clinical outcomes with SOC and some selected regimens among patients diagnosed with stage I-III NSCLC.

DETAILED DESCRIPTION:
The primary objective of this study is to understand the evolution of initial treatment patterns among patients with early-stage (I-III) NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III at initial NSCLC diagnosis
* Aged ≥18 years at first diagnosis of NSCLC
* Timeframe of NSCLC diagnosis:

For DE1: diagnosed with NSCLC during the period between May 1st 2025 and December 31st 2025 For DE2: diagnosed with NSCLC during the period between May 1st 2026 and December 31st 2026 For DE3: diagnosed with NSCLC during the period between May 1st 2027 and December 31st 2027

Exclusion Criteria:

* NSCLC is not the primary cancer diagnosis
* Patients with a recent history of other tumor or concurrent other tumor
* Patients participating in interventional clinical trials at time of initial diagnosis
* Patients with positive pregnancy status at the time of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study will be patients diagnosed with stage I-III NSCLC treated in routine clinical practice with various treatment regimens (e.g., definitive treatment with surgery or radiotherapy, neoadjuvant, adjuvant and perioperative systemic therapies) who meet the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Patterns | Up to 50 months
  Proportion of patients with different treatment regimens
Proportion of unresected patients in SI/II/III | Up to 50 months
  Proportion of patients who are unresected among SI/II/III NSCLC patients enrolled, respectively
CRT rate in USIII | Up to 50 months
  Proportion of patients who have CRT regimen among unresected SIII patients enrolled

SECONDARY OUTCOMES:
Treatment Duration | Up to 50 months
  TKI treatment duration and discontinuation reason in EGFRm patients
  * Duration of treatment
  * Treatment discontinuation (time to discontinuation, and reason for discontinuation)
Patterns of recurrence | Up to 50 months
  Type of recurrence following initial treatment regimen (Loco-regional recurrence, distant recurrence, other)
Guideline adoption rate | Up to 50 months
  Resected EGFRm Stage IB-III
  * Proportion of patients received guideline recommended TKI adjuvant regimen among a. resected EGFRm Stage IB-III patients; b. patients with TKI adjuvant therapy Unresected Stage III
  * Proportion of patients received guideline recommended systemic IO and TKI regimens among patients who received CRT

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified investigators can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/